CLINICAL TRIAL: NCT00591903
Title: Pilot Study to Assess the Proteome in Human Atrial Tissue
Status: Completed | Type: Observational
Sponsor: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Other Study IDs: 999908037; 08-H-N037
Record Dates: First submitted 2007-12-21; First posted 2008-01-11 (Estimated); Last update posted 2017-07-02 (Actual); Status verified 2011-09-23

CONDITIONS: Diabetes; Cardiomyopathy
Keywords: Diabetes and Cardiac Proteomics; Atrial Appendage and Proteomics; Diabetic Cardiomyopathy; Tissue Sample
MeSH Terms: conditions — Diabetes Mellitus; Cardiomyopathies; Diabetic Cardiomyopathies

STUDY DESIGN:
Time Perspective: Prospective

SUMMARY:
The concept of diabetic cardiomyopathy was initially defined more than 30 years ago, as cardiac failure in diabetic subjects in the absence of underlying coronary artery disease. Diabetes is also thought to contribute to earlier stage cardiac systolic dysfunction and/or to isolated diastolic dysfunction, in excess of underlying coronary artery disease and hypertension. More globally, it is recognized that subjects with type 2 diabetes have more extensive cardiovascular disease and a worse outcome for a similar level of disease than non-diabetic subjects. Despite this epidemiological evidence, the biological programming underpinning the myriad presentations of the diabetic heart' are poorly characterized in humans.

Proteomics has emerged as an unbiased technology that enables the measurement of large numbers of steady-state protein levels. The potential to identify a diabetes associated proteomic signature in the heart would be a novel approach to identify putative biological programs altered by the diabetic state.

A portion of the right atrial appendage is removed to insert the cardiac bypass machine cannula in certain cardiothoracic procedures. This tissue is usually discarded, however, we propose that it could be employed to examine whether otherwise similar subjects with and without diabetes have distinct atrial proteomic signatures. This pilot study may provide insight into potential biological pathways that orchestrate the worse cardiac prognosis in type 2 diabetic versus non diabetic control subjects.

DETAILED DESCRIPTION:
The concept of diabetic cardiomyopathy was initially defined more than 30 years ago, as cardiac failure in diabetic subjects in the absence of underlying coronary artery disease. Diabetes is also thought to contribute to earlier stage cardiac systolic dysfunction and/or to isolated diastolic dysfunction, in excess of underlying coronary artery disease and hypertension. More globally, it is recognized that subjects with type 2 diabetes have more extensive cardiovascular disease and a worse outcome for a similar level of disease than non-diabetic subjects. Despite this epidemiological evidence, the biological programming underpinning the myriad presentations of the diabetic heart' are poorly characterized in humans.

Proteomics has emerged as an unbiased technology that enables the measurement of large numbers of steady-state protein levels. The potential to identify a diabetes associated proteomic signature in the heart would be a novel approach to identify putative biological programs altered by the diabetic state.

A portion of the right atrial appendage is removed to insert the cardiac bypass machine cannula in certain cardiothoracic procedures. This tissue is usually discarded, however, we propose that it could be employed to examine whether otherwise similar subjects with and without diabetes have distinct atrial proteomic signatures. This pilot study may provide insight into potential biological pathways that orchestrate the worse cardiac prognosis in type 2 diabetic versus non diabetic control subjects.

ELIGIBILITY:
* INCLUSION CRITERIA:

Subjects must be 18-80 years of age.

Subjects must provide informed, written consent to donate tissue that would otherwise be discarded post-cardiac surgery.

Subjects undergoing elective coronary artery bypass surgery and or aortic valve replacement surgery.

EXCLUSION CRITERIA:

Subjects in atrial fibrillation or having a history of atrial fibrillation in the 2 weeks period prior to surgery.

Use of intravenous anti-arrhythmic therapy.

Subjects unable to give informed consent.

Subjects with a fasting glucose of greater than 110 mg/dl that have not been defined as diabetic.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2007-12-14; Study Completion 2011-09-23

CONTACTS AND LOCATIONS:
Locations (1):
- Suburban Hospital, Bethesda, Maryland, United States

REFERENCES:
- [Background] King H, Aubert RE, Herman WH. Global burden of diabetes, 1995-2025: prevalence, numerical estimates, and projections. Diabetes Care. 1998 Sep;21(9):1414-31. doi: 10.2337/diacare.21.9.1414. PMID 9727886
- [Background] Garcia MJ, McNamara PM, Gordon T, Kannel WB. Morbidity and mortality in diabetics in the Framingham population. Sixteen year follow-up study. Diabetes. 1974 Feb;23(2):105-11. doi: 10.2337/diab.23.2.105. No abstract available. PMID 4359625
- [Background] Rubler S, Dlugash J, Yuceoglu YZ, Kumral T, Branwood AW, Grishman A. New type of cardiomyopathy associated with diabetic glomerulosclerosis. Am J Cardiol. 1972 Nov 8;30(6):595-602. doi: 10.1016/0002-9149(72)90595-4. No abstract available. PMID 4263660